CLINICAL TRIAL: NCT06433011
Title: The RAPID - PE Study: RESCUE Advanced Protocol Without ICU Stay and no Lytic Drip - for the Treatment of Pulmonary Embolism
Brief Title: The RAPID - PE Study: RESCUE Advanced Protocol for the Treatment of Pulmonary Embolism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thrombolex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THRO-CLIN-2024-01
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Catheter Directed Therapy
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Pulse Spray and Infusion of r-tPA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- BEC Treatment (Experimental): The Bashir™ Endovascular Catheter is a device intended for the localized infusion of therapeutic agents into the pulmonary artery.
  Interventions: Device: The Bashir™ Endovascular Catheter; Drug: r-tPA

INTERVENTIONS:
Device: The Bashir™ Endovascular Catheter — The Bashir™ Endovascular Catheter is a device intended for the localized infusion of therapeutic agents into the pulmonary artery and peripheral vasculature.
Drug: r-tPA — Pulse spray and infusion

SUMMARY:
To demonstrate the efficacy and safety of the 8F BASHIR™ .035 Endovascular Catheter and the 8F BASHIR™ S-B .035 Endovascular Catheter for the administration of pharmaco-mechanical catheter directed therapy using pulse sprays of r-tPA into the pulmonary arteries for the treatment of intermediate risk pulmonary embolism (PE).

DETAILED DESCRIPTION:
The BASHIR™ .035 Endovascular Catheter (BEC) and the BEC Short Basket .035 (S-B) are devices intended for the localized infusion of therapeutic agents into the pulmonary artery and peripheral vasculature. The distal infusion segment of the device contains an expandable radial array of conduits with a total of 48 laser drilled orifices used for the delivery of the therapeutic agents at multiple cross-sectional points of the target vessel location. The infusion segment can be expanded and collapsed by the actuator (slider) located on the handle at the proximal end of the device. The infusion line connector is also located on the handle. The difference between the BEC .035 and the BEC S-B.035 is solely in the length of the basket. In its unexpanded state, the basket of the BEC .035 is 12.5cm long and the BEC S-B .035 basket is 10cm long. The choice of device used will be at the physician's discretion based on the patient's anatomy.

ELIGIBILITY:
Inclusion Criteria

1. Willing and able to provide informed consent;
2. PE symptom duration ≤ 15 days;
3. Filling defect in at least one major lobar pulmonary artery as determined by CTA;
4. Patient is diagnosed with intermediate risk PE;
5. RV/LV diameter ratio ≥ 0.9 by CTA, as determined by investigative site;
6. Willing and able to comply with all study procedures and 7-day and 30-day telephone follow-up visit.

Exclusion Criteria:

1. Previous history of stroke with residual hemiplegia;
2. Major surgery ≤ 10 days prior to inclusion in the study;
3. Platelet count < 100,000/μL;
4. Pulmonary thrombectomy within the previous 4 days;
5. Uncontrolled hypertension defined as systolic blood pressure >180 mm Hg and/or diastolic blood pressure >110 mm Hg at the time of the procedure;
6. Administration of thrombolytic agents within the previous 4 days;
7. Absolute contraindication to anticoagulation;
8. Clinician deems high-risk for catastrophic bleeding;
9. Pregnancy;
10. Any vasopressor or inotropic support;
11. Cardiac arrest (including pulseless electrical activity (PEA) and asystole) requiring active cardiopulmonary resuscitation (CPR) during this hospitalization at treating institution and/or referring institution;
12. Planning to administer r-tPA by infusion after the r-tPA is administered by pulse sprays;
13. Currently participating in another study;
14. In the opinion of the investigator, the subject is not a suitable candidate for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-06-25 (Estimated); Primary Completion 2027-06-25 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Death from any cause or hemodynamic decompensation (or collapse) | Procedure through 7-day follow-up
  Observe death from any cause or hemodynamic decompensation (or collapse) through 7-day follow-up, defined as need for cardiopulmonary resuscitation; or
  1. SBP < 90 mmHg for at least 15 minutes; or
  2. drop in SBP by at least 40 mmHg for at least 15 minutes with signs of end-organ hypoperfusion (cold extremities or low urinary output < 30 mL/h or mental confusion); or
  3. need for catecholamine administration to maintain adequate organ perfusion and a SBP > 90 mmHg (including dopamine at the rate of > 5 micrograms / kg per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Mifek, Study Director — Thrombolex, Inc.

IPD SHARING:
Plan to Share IPD: No